CLINICAL TRIAL: NCT03458156
Title: Clinical Study of Umbilical Cord Mesenchymal Stem Cell Transplantation for Lupus Nephritis
Brief Title: Umbilical Cord Mesenchymal Stem Cell Transplantation for Lupus Nephritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Liu Jing, Chief Physician, The First Affiliated Hospital of Dalian Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DalianMU_JL_002
Record Dates: First submitted 2018-02-07; First posted 2018-03-08 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SLE group (Experimental): The patients will be assigned to systemic lupus erythematosus (SLE) group, receiving umbilical cord mesenchymal stem cell transplantation.
  Interventions: Biological: SLE group
- LN group (Experimental): The patients will be assigned to lupus nephritis (LN) group, receiving umbilical cord mesenchymal stem cell transplantation.
  Interventions: Biological: LN group
- the control group (Experimental): The patients will be assigned to the control group.
  Interventions: Other: the control group

INTERVENTIONS:
Biological: SLE group — The patients will be assigned to systemic lupus erythematosus (SLE) group, receiving umbilical cord mesenchymal stem cell transplantation.
  Arms: SLE group
Biological: LN group — The patients will be assigned to lupus nephritis (LN) group, receiving umbilical cord mesenchymal stem cell transplantation.
  Arms: LN group
Other: the control group — The patients will be assigned to the control group.
  Arms: the control group

SUMMARY:
To investigate the safety and efficacy of umbilical cord mesenchymal stem cell transplantation in patients with systemic lupus erythematosus (SLE) and lupus nephritis (LN).

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a multisystem autoimmune disease. Lupus nephritis (LN) is one of the most serious complications of SLE. The current clinical treatments of LN mainly include steroids and immunosuppressive drugs, but drug side effects are obvious.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the 1997 American College of Rheumatology (ACR) classification criteria of SLE.
* age 18-60 years.
* of either sex and of any ethnicity.
* Lupus nephritis (LN) group: (1) Receiving more than 6 months of regular treatment, 24-hour urine protein ≥ 1.0 g, serum creatinine ≥1.5 mg/dL; (2) renal biopsy: class III, IV or V LN included, and class VI excluded.
* After conventional treatment (glucocorticoid therapy and immunosuppressive drugs) prior to grouping, SLEDAI scores ≥ 10.
* Receiving 12 months of treatment while using birth control.
* Provision of informed consent.

Exclusion Criteria:

* Poor blood pressure control by drug treatment (≥ 160/100 mmHg)
* Abnormal hepatic function (a 3-fold increase in alanine aminotransferase level relative to normal liver).
* Renal failure (glomerular filtration rate < 15 mL/min/1.73 m2).
* Severe heart and lung failure, or injury to other important organs
* Uncontrollable infection.
* Having not taken biological agents for 6 months.
* Pregnant or lactating women, or those women who are trying to get pregnant or those men who are trying to make their partners pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-09 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
SLEDAI-2000 score | changes of month 3, month 6, month 9 and month 12 after treatment
  The SLEDAI 2000 is a novel index that measures ≥ 50% in each of the 24 descriptors of SLEDAI-2K and generates a total score reflecting disease activity overall.

SECONDARY OUTCOMES:
BILAG-2004 score | changes of month 3, month 6, month 9 and month 12 after treatment
  The BILAG-2004 is a comprehensive composite clinical index that has been recently validated for the assessment of systemic lupus erythematosus (SLE) disease activity. This index is based on the Classic BILAG index and has many similarities with its predecessor: it is based on the principle of the physician's intention to treat, has transitional property that captures changing severity of clinical manifestations and has a similar ordinal scale scoring system. However, it has nine systems and many of the changes (from the Classic BILAG index) are in the items, glossary and scoring scheme. As with the Classic BILAG index, the individual system scores were not intended to be summated into a global score.
Health Assessment Questionnaire (HAQ) score | changes of month 3, month 6, month 9 and month 12 after treatment
  The Health Assessment Questionnaire (HAQ) has played an influential role in establishing health outcome assessment as a quantifiable set of reliable, valid and responsive hard data points. The HAQ is based on five patient-centered dimensions: disability, pain, medication effects, costs of care, and mortality. It has been validated by mail, in the office, by telephone, and by comparison with paraprofessional and physician judgments as a reliable instrument, and has been significantly correlated with other PRO instruments. Typically, one of two HAQ versions is used: the Full HAQ, which assesses all five dimensions, and the Short or 2-page HAQ, which contains only the HAQ disability index (HAQ-DI) and the HAQ's patient global and pain visual analog scales (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Liu Jing, Ph.D, Principal Investigator — The First Affiliated Hospital of Dalian Medical University

IPD SHARING:
Plan to Share IPD: Undecided